CLINICAL TRIAL: NCT01809249
Title: Causes of Disqualification of Egyptian Potential Living Liver Donors
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Lecturer of Tropical Medicine, Ain Shams University
Other Study IDs: Donar Safety
Record Dates: First submitted 2013-03-09; First posted 2013-03-12 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Donors Safety
Keywords: Living donor liver transplantation; Donar safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Due to absence of Deceased-donors in Egypt, Living-donor liver transplantation (LDLT) has emerged as an option to the traditional deceased-donor transplantation procedure. But there is an essential risk related to liver resection for healthy donors.

DETAILED DESCRIPTION:
The aim of this work is to identify and analyze the causes of disqualification of potential Egyptian living liver-donors in a University based liver transplant program

ELIGIBILITY:
Inclusion Criteria:

* All potential living liver donors in the period from June 2010 to June 2012

  1. Age between 18 and 50 years
  2. Relationship within 3rd degree of consanguinity with recipient or spouse.
  3. The donor-recipient pair must be blood group compatible.
  4. An informed consent should be obtained.

Exclusion Criteria:

* Patients with nknown mrsdical or surgical history that interfere with donation

  * Underlying medical condition (diabetes, cardiopulmonary disease, etc.).
  * ABO incompatibility

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: potential living liver donors
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
causes of disqualification of potential Egyptian living liver-donors | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Center For Organ Transplantation (ASCOT),Ain Shams university, Cairo, Egypt